CLINICAL TRIAL: NCT06794944
Title: Use of Fidaxomicin Compared to Vancomycin for Decolonization of C. Difficile in Patients With Inflammatory Bowel Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jessica Ravikoff Allegretti, Jessica Ravikoff Allegretti, MD, MPH, FACG, AGAF, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P000187
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Bowel Disease (IBD); Clostridioides Difficile Infection
Keywords: C. difficile; Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Clostridium Infections; Colitis, Ulcerative | interventions — Vancomycin; Fidaxomicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vancomycin (Active Comparator): Vancomycin is glycopeptide antibiotic that has broad gram-positive coverage. The current approved dose is 125mg PO every 6 hours for 10 days. Appropriate dosing and tolerance of vancomycin is well defined in both healthy and hospitalized populations, as it is already approved and indicated by the FDA for use in treating C. difficile infection.
  Interventions: Drug: Vancomycin (POC)
- Fidaxomicin (Active Comparator): Fidaxomicin is a macrolide antibiotic. It is narrow spectrum with potent bactericidal activity specifically against C. difficile. The approved dose is 200mg PO twice daily for 10 days. Appropriate dosing and tolerance of fidaxomicin is well defined in both healthy and hospitalized populations, as it is already approved and indicated by the FDA for use in treating C. difficile infection.
  Interventions: Drug: Fidaxomicin

INTERVENTIONS:
Drug: Vancomycin (POC) — Vancomycin is glycopeptide antibiotic that has broad gram-positive coverage. Patients will receive 125mg PO every 6 hours for 10 days.
  Arms: Vancomycin
Drug: Fidaxomicin — Fidaxomicin is a macrolide antibiotic. It is narrow spectrum with potent bactericidal activity specifically against C. difficile. Patients will receive 200mg PO twice daily for 10 days.
  Arms: Fidaxomicin

SUMMARY:
This is a randomized, double-blind study to assess the safety and efficacy of fidaxomicin compared to vancomycin for decolonization of C. difficile in IBD patients. A total of 60 patients who meet eligibility criteria will be randomized 1:1 to either the fidaxomicin or vancomycin arm. The vancomycin arm will receive a dose of 125 mg PO q 6 hours for 10 days. The fidaxomicin arm will receive 200 mg PO BID for 10 days. In order to ensure blinding, both antibiotics will be concealed in opaque 00 capsule shells. In addition, those in the fidaxomicin arm will receive 2 placebo capsules so that all participants will receive 4 capsules daily for 10 days. Microbiome assessment and C. difficile testing will be performed at baseline, day 5, day 10, and weeks 4, 8, and 26.

DETAILED DESCRIPTION:
This randomized, double-blind trial will assess the ability of fidaxomicin compared to vancomycin to decolonize C. difficile in the IBD patient population.

Participants who meet eligibility criteria will be randomized 1:1 to either vancomycin or fidaxomicin treatment. The vancomycin arm will receive a dose of 125 mg PO q 6 hours for 10 days. The fidaxomicin arm will receive 200 mg PO BID for 10 days. In order to ensure blinding both antibiotics will be concealed in opaque 00 capsule shells. In addition, those in the fidaxomicin arm will receive 2 placebo capsules so that all participants will receive 4 capsules daily for 10 days. Participants will end dosing after 10 days, but monitoring will continue to week 8. Both participants and study team will be blinded to treatment arm allocation.

Participants will be assessed through week 8 for the primary outcome, decolonization. Safety and tolerability outcomes will be assessed through week 8. In addition, secondary efficacy outcomes including IBD disease activity and development of CDI will be evaluated at week 8 and week 26. Participants will also be followed through week 26 for long-term safety, efficacy, and clinical outcomes. Disease activity and symptoms will be recorded from time of informed consent through to the week 26 trial visit. Stool samples for biomarker assessments and C. difficile testing will be collected at scheduled trial visits per Schedule of Assessments.

The primary outcome, decolonization of C. Difficile at week 8, will be confirmed via stool sampling. Additional C. difficile testing will be done at week 26.

Participants that experience intolerable adverse events will be withdrawn from the study and will be considered treatment failures. Additional subjects may be enrolled to obtain 60 patients with week 8 data.

The study will enroll approximately 60 adult participants at a single center.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Male or female > 18 years of age.
3. IBD diagnosis (CD, UC or indeterminant Colitis will be permitted.)
4. Presenting for outpatient colonoscopy for any indication.

Exclusion Criteria:

1. Unable to provide consent.
2. Patients with previous colectomy, ostomy, J-pouch, or previous colon surgery (excluding appendectomy.)
3. Unable to complete study procedures.
4. Chronic use of antibiotics.
5. Inability or unwillingness to swallow capsules.
6. Allergy or sensitivity to vancomycin, fidaxomicin, or microcrystalline cellulose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
C. difficile decolonization | 8 weeks
  Absence of C. difficile via PCR in Week 8 stool sample
Safety and tolerability | 8 weeks
  Subject incidence of treatment-emergent adverse events (including treatment-emergent adverse events for clinically significant changes in laboratory parameters and vital signs)

SECONDARY OUTCOMES:
Biomass of C. difficile | 8 weeks
  Change in stool C. difficile biomass in patients at week 8 by quantitative culture and qPCR
Long-term effect of C. difficile decolonization on IBD clinical outcomes | 26 weeks
  Change in IBD clinical scores from baseline at week 8 and week 26. IBD clinical scores are used to assess IBD patient symptoms. The assessments are separated between scores for Ulcerative Colitis (UC) and Crohn's Disease (CD). The Harvey Bradshaw Index (HBI) is a clinical assessment for IBD patients with Crohn's disease while Partial Mayo Score is a clinical assessment for Ulcerative Colitis. The scores will be collected at study visit in form of a survey. The HBI score can vary but a score above 8 or 9 is considered severe disease activity. The Partial Mayo Score can range from 0 to 9 and a score above 7 is considered severe disease activity. A decrease in score from baseline to follow-up timepoints is indicative of improved IBD patient symptoms. A decrease in score from baseline to follow-up timepoints is indicative of improved IBD patient symptoms.
C. difficile infection surveillance | 26 weeks
  Incidence of patients developing CDI through Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Allegretti, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No